CLINICAL TRIAL: NCT05818111
Title: Comparison of Different Volume of Steroid Hydrodilatation in Treating Patients With Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-12-001B
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-12

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis
MeSH Terms: conditions — Bursitis | interventions — Steroids; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low volume hydrodilatation (Experimental): patient received ultrasound-guided low volume steroid hydrodilatation (4cc shincort + 4cc 2% xylocaine +2cc normal saline)
  Interventions: Drug: steroid; Drug: Xylocaine 2 % Injectable Solution; Drug: Normal saline 2cc
- high volume hydrodilatation (Active Comparator): patient received ultrasound-guided high volume steroid hydrodilatation (4cc shincort + 4cc 2% xylocaine +12cc normal saline)
  Interventions: Drug: steroid; Drug: Xylocaine 2 % Injectable Solution; Drug: normal saline 12cc

INTERVENTIONS:
Drug: steroid — triamcinolone 40mg 4cc
Drug: Xylocaine 2 % Injectable Solution — xylocaine 2% 4cc
Drug: Normal saline 2cc — normal saline 2cc
  Arms: low volume hydrodilatation
Drug: normal saline 12cc — normal saline 12cc
  Arms: high volume hydrodilatation

SUMMARY:
This study was conducted to compare the efficacy of low volume steroid hydrodilatation with high volume steroid hydrodilatation under ultrasonographic guidance for treating adhesive capsulitis

DETAILED DESCRIPTION:
adhesive capsulitis is a common cause of shoulder pain, and the efficacy of most interventions is limited. This study was conducted to compare the efficacy of low volume steroid hydrodilatation with high volume steroid hydrodilatation under ultrasonographic guidance for treating adhesive capsulitis Design: a prospective, double-blinded, randomized, clinical trial

Patient and methods:

Patients with adhesive capsulitis for at least 3 months were enrolled and randomly allocated into group 1 (10cc steroid hydrodilatation under ultrasonographic guidance ) and group 2 (20cc steroid hydrodilatation). The patients were evaluated before treatment and were reevaluated 0, 6, and 12 weeks after the beginning of the treatment. Outcomes measures included a pain scale (visual analog scale), range of motion, Shoulder Pain And Disability Index

ELIGIBILITY:
Inclusion Criteria:

1) age 35-65 years (to prevent the inclusion of patients with secondary AC), 2) onset of shoulder stiffness since over a month, and 3) limitation in the passive range of motion (ROM) over 30° when compared with the contralateral side in at least two of these three movements: forward flexion, abduction, or external rotation.

Exclusion Criteria:

1. ultrasound findings of rotator cuff tears, 2) plain radiography findings of significant glenohumeral joint arthritis, 3) accompanying cervical radiculopathy, 4) systemic inflammatory joint disease, 5) intraarticular injection into the glenohumeral joint within the past 3 months, 6) history of surgery on the affected shoulders, 7) regular use of systemic non-steroidal anti-inflammatory drugs or corticosteroids, and 8) allergy to corticosteroid or lidocaine.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
change in visual analog scale visual analog scale | at 6, 12 wk
  visual analog scale

SECONDARY OUTCOMES:
change in glenohumeral joint range of motion | at 6, 12 wk
  Shoulder flexion, abduction, external rotation and internal rotation were measured with goniometer with patient in supine position.
change in Shoulder Pain And disability index | at 6, 12 wk
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
change in pain intensity | at 6, 12 wk
  pain intensity was measured by visual analog scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan